CLINICAL TRIAL: NCT02995083
Title: Corticosteriods vs. Saline vs. Air Placebo Intra-articular Injections for Knee Osteoarthritis: A Single Blinded Prospective Randomized Trial
Brief Title: Intra-articular Injections for Knee Osteoarthritis: A Single Blinded Prospective Randomized Trial
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study deemed not feasible
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Mukesh Ahuja, Certified Principal Investigator, Research Administrator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16090902
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Symptomatic Osteoarthritis of the Knee
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone Acetate; Lidocaine; Adrenal Cortex Hormones; Saline Solution; Sodium Chloride; Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Knee injection with corticosteroids (Active Comparator): Using clinically accepted methods, subjects will undergo a palpation guided injection of corticosteroids into the knee joint. Subjects will then return for follow-up visit at 12 weeks for a physical exam of the knee. Patients will fill out questionnaires online at 1, 6, 12 and 24 weeks.
  Interventions: Drug: 40 mg Depo-Medrol in 1 ml, 9 ml of 1% lidocaine
- Knee injection with saline (Placebo Comparator): Using clinically accepted methods, subjects will undergo a palpation guided injection of saline into the knee joint. Subjects will then return for follow-up visit at 12 weeks for a physical exam of the knee. Patients will fill out questionnaires online at 1, 6, 12 and 24 weeks.
  Interventions: Drug: Normal Saline 10 ml
- Knee injection with air (Sham Comparator): Using clinically accepted methods, subjects will undergo a palpation guided injection of air into the knee joint. Subjects will then return for follow-up visit at 12 weeks for a physical exam of the knee. Patients will fill out questionnaires online at 1, 6, 12 and 24 weeks.
  Interventions: Drug: Air 10 ml

INTERVENTIONS:
Drug: 40 mg Depo-Medrol in 1 ml, 9 ml of 1% lidocaine — Patients will receive an ultrasound guided intra-articular injection of 40 mg Depo-Medrol in 1 ml, 9 ml of 1% lidocaine
  Other Names: Corticosteroid
  Arms: Knee injection with corticosteroids
Drug: Normal Saline 10 ml — Patients will receive an ultrasound guided intra-articular injection of Normal Saline 10 ml
  Other Names: Saline
  Arms: Knee injection with saline
Drug: Air 10 ml — Patients will receive an ultrasound guided intra-articular injection of Air 10 ml
  Other Names: Air
  Arms: Knee injection with air

SUMMARY:
To investigate the clinical benefit of intra-articular injections of saline in patients with symptomatic osteoarthritis of the knee and compare the clinical response of saline to the current standard treatment with corticosteroids and an air injection placebo.

DETAILED DESCRIPTION:
As non-surgical treatments of OA are essential, multiple trials have been done to compare standard of care IA injection therapies to more novel injection treatments, with many of these trials using saline as the control arm. The purpose of using a control arm is to attempt to eliminate placebo effect and help distinguish the true effectiveness of a therapy. There has been controversy over the clinical effect of saline in treating OA with some arguing that saline may have some clinical benefit. If this is true, it could allow for the true effect of standard of care therapies to appear diminished when compared to saline as a placebo. A recent meta analysis looked at the use of saline as a placebo in 38 randomized control trials to determine if intra-articular saline injections for knee OA had a clinical effect. The study found that IA injections of saline significantly improved short-term knee pain in 32 of the studies which involved 1705 patients, p <0.001, and long-term pain was significantly decreased in 19 of the studies involving 1445 patients, p <0.001. It is essential to empirically determine if saline has a clinical effect due to the role it plays as a placebo in many clinical studies of the management of OA with intra-articular injections.

Objective: To investigate the clinical benefit of intra-articular injections of saline in patients with symptomatic osteoarthritis of the knee and compare the clinical response of saline to the current standard treatment with corticosteroids and an air injection placebo.

Study Design: Prospective, single-blinded, randomized, clinical study. Patients will be randomized into three treatment arms in a 1:1:1 fashion with approximately 50 patients in the saline arm, 50 patients in the corticosteroid arm, and 50 patients in the placebo arm.

Null Hypothesis: Clinical knee outcomes of subjects following one intra-articular knee injection of air will be similar to one intra-articular knee injection of saline or corticosteroid for symptomatic patients diagnosed with knee OA.

Statistical Assumptions: Power Analysis

Investigational Arm: 10 ml Saline (Normal Saline)

Control Arm: 1 ml of 40 mg corticosteroid in 9 ml 1% lidocaine (Depo-medrol, Pfizer, New York, New York), 10 ml air (placebo)

Primary Efficacy Endpoint: The primary efficacy endpoint is the mean change in the WOMAC Index score 12 weeks after first injection with regards to baseline score.

Secondary Efficacy Secondary efficacy endpoints include the change in the full Endpoints: WOMAC Index, KOOS, Lysholm, IKDC, VAS, SF-12 and use of rescue medication (steroid at 12 weeks).

Enrollment: Prospective, randomized, clinical study designed to evaluate 150 subjects. All enrolled subjects will have a pre-procedure visit, one treatment visit, and follow-up visits at week 6 and week 12 if they require a rescue injection and will fill out patient reported outcome measures at 1, 6, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be between the ages of 18 and 80
2. Informed consent has been obtained from the patient
3. The patient must have diagnosed symptomatic osteoarthritis of the tibio-femoral or patello-femoral compartment of the target knee for at least 1 month
4. The patient has moderate-to-severe knee pain reflected by an average visual analogue scale (VAS) score of 4 or greater (out of a possible 10) over the previous 7 days.
5. Radiographic imaging must show grade II-III osteoarthritis on the Kellgren & Lawrence Scale.
6. Patients may have bilateral osteoarthritis but only patients with unilateral symptoms may be included.

Exclusion Criteria:

1. Knee instability
2. A score less than 4 (out of a possible 10) on their intake VAS
3. Major axial deviation (>5º valgus or varus deviation as evidenced on a standard of care x-ray.
4. Previous surgery at the target knee < 6 months.
5. Symptomatic osteoarthritis of the contralateral knee or any other joint.
6. Systemic or intra articular injection to any joint with corticosteroids within 6 months prior to screening
7. Previous joint injection of any type in the past 6 months
8. Systemic conditions that could interfere with outcome such as Rheumatoid arthritis, coagulopathy, and anemia.
9. Allergy to any of the injected substances.
10. Any patient unable to cease NSAID usage (other than low dose aspirin) due to unrelated condition.
11. Cognitive impairment or unable to provide informed consent
12. Recent knee trauma with violation of the intra-articular bone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in Western Ontario and McMaster Universities Arthritis Index score (WOMAC) | 12 weeks after injection
  Mean change in the WOMAC Index score from baseline score

SECONDARY OUTCOMES:
Mean change in Knee injury and Osteoarthritis Outcome Score (KOOS) | 12 weeks after injection
  Mean change in the KOOS from baseline score
Mean change in International Knee Documentation Committee (IKDC) score | 12 weeks after injection
  Mean change in IKDC from baseline score
Mean change in Visual Analogue Scale (VAS) | 12 weeks after injection
  Mean change in VAS from baseline score
Mean change in Short Form 12 (SF-12) score | 12 weeks after injection
  Mean change in SF-12 from baseline score
Mean change in The Lysholm Knee score | 12 weeks after injection
  Mean change in The Lysholm Knee score from baseline score
Mean change in use of rescue medication | 12 weeks after injection
  Use of anti-inflammatory, analgesics, and rescue corticosteroid injection. Number of pills taken each day. This will be collected via survey. If the medical examiner feels that the patient is continuing to do poorly and they did not receive the steroid injection intervention, then they will be offered a rescue corticosteroid injection at 12 weeks. The number of patients who do not initially receive a corticosteroid injection and require a rescue corticosteroid injection at 12 weeks will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil N Verma, MD, Principal Investigator — Midwest Orthopaedics at Rush University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Altman RD, Devji T, Bhandari M, Fierlinger A, Niazi F, Christensen R. Clinical benefit of intra-articular saline as a comparator in clinical trials of knee osteoarthritis treatments: A systematic review and meta-analysis of randomized trials. Semin Arthritis Rheum. 2016 Oct;46(2):151-159. doi: 10.1016/j.semarthrit.2016.04.003. Epub 2016 Apr 27. PMID 27238876
- [Background] Williams VJ, Piva SR, Irrgang JJ, Crossley C, Fitzgerald GK. Comparison of reliability and responsiveness of patient-reported clinical outcome measures in knee osteoarthritis rehabilitation. J Orthop Sports Phys Ther. 2012 Aug;42(8):716-23. doi: 10.2519/jospt.2012.4038. Epub 2012 Mar 8. PMID 22402677
- [Background] Kim J, Seo BS. How to calculate sample size and why. Clin Orthop Surg. 2013 Sep;5(3):235-42. doi: 10.4055/cios.2013.5.3.235. Epub 2013 Aug 20. PMID 24009911
- [Background] Zhang W, Robertson J, Jones AC, Dieppe PA, Doherty M. The placebo effect and its determinants in osteoarthritis: meta-analysis of randomised controlled trials. Ann Rheum Dis. 2008 Dec;67(12):1716-23. doi: 10.1136/ard.2008.092015. Epub 2008 Jun 9. PMID 18541604
- [Background] Eker HE, Cok OY, Aribogan A, Arslan G. The efficacy of intra-articular lidocaine administration in chronic knee pain due to osteoarthritis: A randomized, double-blind, controlled study. Anaesth Crit Care Pain Med. 2017 Apr;36(2):109-114. doi: 10.1016/j.accpm.2016.05.003. Epub 2016 Jul 30. PMID 27485803